CLINICAL TRIAL: NCT04039568
Title: Meditation Versus Education for Improving Depression in Chronic Pain, a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Lunenfeld Tanenbaum Research Institute (Other); Rivlin Medical Group (Unknown); The Art of Living Foundation (Other); Canadian Mental Health Association (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Ross Upshur, Principal Investigator, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EO1-162072; EO1-162072 (Other Grant/Funding Number: Canadian Institute of Health Research)
Record Dates: First submitted 2019-07-15; First posted 2019-07-31 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain; Depression
Keywords: Opioid Therapy; Sahaj Samadhi Meditation; Health Enhancement Program
MeSH Terms: conditions — Chronic Pain; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Control Group (Active Comparator): Ten to fifteen participants in the HEP arm will participate in the program for 4 consecutive days (2hrs/day) in the 1st week, followed by 75 min/week reinforcement sessions for 11 weeks.
  The Health-Enhancement Program (HEP) was designed and used as a manualized active control in meditation-based intervention trials. HEP controls for several non-specific factors found in a meditation groups, including: group support and morale, behavioural activation, reduction of stigma, facilitator attention, treatment duration, and time spent on at-home practice. HEP is tailored to be structurally equivalent to SSM with similar-sized groups, meeting schedule, total contact hours, amount of home practice and encouragement to keep practice logs.
  Interventions: Behavioral: Health Enhancement Program (HEP)
- Intervention Group (Experimental): Ten to fifteen participants in the SSM arm will be trained for 4 consecutive days (2hrs/day) in the 1st week, followed by 75 min/week reinforcement sessions for 11 weeks.
  This standardized, manualized therapy will be delivered by certified meditation instructors. On day 1, participants will learn the nature of meditation, and then undergo personal guided meditation. Training on days 2-4 includes understanding the nature of the mind and the thoughts arising from it, guided meditations by the instructor, and a discussion of meditation processes. Weekly 75 min reinforcement sessions will include 20 minutes of guided meditation practice, and then focus on participants' experiences with meditation during the week, additional observations, and a review of relevant knowledge to support their home practice. Participants will also be encouraged to practice twice daily at home for 20 minutes per session.
  Interventions: Behavioral: Sahaj Samadhi Meditation (SSM)

INTERVENTIONS:
Behavioral: Health Enhancement Program (HEP) — This is the active control group of the study, where participants will be educated on health promotion, healthy diet, music, and exercise, but do not learn breathing techniques, or meditation.
  Arms: Active Control Group
Behavioral: Sahaj Samadhi Meditation (SSM) — This is the experimental arm of the study, where participants will be trained in a form of meditation that may improve depressive symptoms.
  Arms: Intervention Group

SUMMARY:
In this study two possible treatment options available for depression and chronic pain will be explored. Both of these treatments will be offered through online group video calls, which could translate to cost-savings for the health care system. The two treatment options are:

1. The Health Enhancement Program (HEP). Designed to give participants information and guidance on how to lead a healthy lifestyle, which could be beneficial in treating depression.
2. Sahaj Samadhi Meditation (SSM). A unique and easy-to-learn meditation technique that reduces stress and provides deep relaxation which could be beneficial in treating depression.

This study will use a hybrid type 1 evaluation design that primarily focuses on a single-site, single-blinded (investigator, and clinician), 12-week randomized controlled trial (RCT) comparing SSM (n=80) versus HEP (n=80) in 160 adults with depression and chronic pain. Participants will be blinded to the treatment hypothesis while investigators, raters and treating clinicians will be additionally blinded to the intervention. Evaluations of depression (PHQ-9), pain symptoms (BPI), quality of life (SF-36), and opioid use will be collected at baseline, intervention completion (12 week), and at 24 week follow-up. An implementation evaluation will draw from four key study populations: (1) the participants of the RCT; (2) the expert meditation instructors facilitating the intervention; (3) the site staff and investigators involved in supporting the logistics of the intervention arm of the RCT.

DETAILED DESCRIPTION:
OBJECTIVES To determine whether depressive symptoms, pain severity, function, quality of life, as well as opioid use can be affected by a lifestyle intervention program in depression and chronic pain. To evaluate the implementation of the program at Rivlin Medical Group (RMG) chronic pain clinic, and to understand how the SSM intervention can be translated to other settings.

RCT RECRUITMENT AND CONSENT Adults with chronic pain and depression will be recruited from one of seven sites: 1) the Rivlin Medical Group Clinic, 2) Mount Sinai Academic Family Health Team, Sinai Health, 3) TAPMI hub programs at Women's College Hospital 4) Academic Family Health Team, St. Michael's Hospital, 5) the Rehabilitation Pain Service, University Health Network, 6) the Canadian Memorial Chiropractic College sites, and 6) South East Toronto Family Health Team, Michael Garron Hospita. Recruitment materials (brochure, poster, website) will also be shared at local independent non-hospital sites and in online spaces. Patients will be introduced to the study and connected with study staff. All potential participants will be provided with a consent form and given a minimum of 24 hours to consider participation. After this time, informed consent will be obtained from those interested in participating and they will be screened for eligibility by study staff.

STUDY INTERVENTIONS This study is a 12-week, randomized controlled trial seeking to recruit 160 participants with depression and chronic pain. The SSM intervention will be offered by trained and certified teachers from the Art of Living Foundation. The HEP intervention will be offered by a trained Nurse Practitioner, Social Worker, Psychologist, Occupational Therapist or other qualified healthcare professional. Raters, clinicians, and care providers will be blind to participant study condition.

DATA COLLECTION Participants will be screened for eligibility using the Patient Health Questionnaire (PHQ-9) and Mini International Neuropsychiatric Interview Screen and Standard 7.0.2 (MINI). The primary outcome (depression) will be evaluated using the PHQ-9. The secondary outcome (pain severity and pain-related function) will be evaluated using the Brief Pain Inventory (BPI. Exploratory outcomes (health related quality of life, and opioid use) will be evaluated using the Short-form 36 (SF-36), and a medication log, respectively. Measures of primary and secondary outcomes will be administered at all 3 assessment sessions and are described below.

At the baseline assessment the following information will be collected:

i. Demographics survey that will collect information on age, partial Date of Birth (DOB), gender, ethnic background, employment status, housing type, highest level of education achieved, smoking, caffeine intake, drug and alcohol use, duration of pain and pain diagnosis. Participants will also be asked about their psychiatric history including age of first contact with services for mental illness (and which illness), history of hospital admissions and the number of episodes of depression; ii. PHQ-9; iii. BPI scale; iv. SF-36; v. Medication names, dosages, dosages per day, total daily dosage, and reason for use will be recorded, including vitamins and over-the-counter (OTC) medications; vi. Psychology Intake Form.

During the 12 week and 6 month assessment the following questionnaires and measurements will be completed:

i. PHQ-9; ii. BPI scale; iii. SF-36; iv. Medication names and doses will be collected and the recordings for opioids will be converted to total daily morphine equivalents using standardized conversion tables.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. 2. Significant depressive symptomology (PHQ-9 score ≥10);
3. Chronic pain (pain ≥3 months duration in any body region, by self-report);
4. Be willing and able to attend all 4 training sessions of SSM/HEP and 75% of follow-up sessions;
5. Understanding of English language (spoken and written);
6. Able to sit for 20-25 minutes without significant discomfort;
7. Regular access to internet and ability to participate in video calls

Exclusion Criteria:

1. Other major psychiatric conditions including substance use disorder, psychosis and cognitive impairment as excluded by the Mini-International Neuropsychiatric Interview (MINI) Screening and Standard tool; severe depression (PHQ-9 ≥20) and risk of imminent suicide as per MINI and/or PHQ-9;
2. Non-correctable, clinically significant sensory impairment;
3. Acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months;
4. A terminal medical diagnosis with prognosis of less than 12 months;
5. Currently practising any form of mind-body intervention;
6. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Health and Depression Symptomology | Baseline (Week 0), Follow-up 1 (Study completion; Week 12-13), Follow-up 2 (Week 24)
  The Patient Health Questionnaire (PHQ-9) is a well-validated and widely used self-report scale used in depression and chronic pain clinical care and research. Reduction in a continuous outcome score is a more sensitive test viz a viz percent reduction in scores which has been reported in some depression studies.

SECONDARY OUTCOMES:
Change in Pain Severity and pain-related function | Baseline (Week 0), Follow-up 1 (Study completion; Week 12-13), Follow-up 2 (Week 24)
  The Brief Pain Inventory (BPI) is a validated self-report scale used in pain trials and clinical pain practice and is a core outcome measure per the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) recommendations. Two independent measures are included: pain severity and pain interference with function - both are clinically relevant outcomes.

OTHER OUTCOMES:
Change in Medication Information | Baseline (Week 0), Follow-up 1 (Study completion; Week 12-13), Follow-up 2 (Week 24)
  Opioid dose will be collected via patient log is the most common measure of opioid use in clinical research trials as per our current review of multidisciplinary care for opioid tapering. Given that patients are on a variety of distinct opioids and that single patients may be on >1 formulation, there is a need for common reporting as provided by morphine equivalent doses. Other prescription medications will also be recorded
Change in Health-Related Quality of Life | Baseline (Week 0), Follow-up 1 (Study completion; Week 12-13), Follow-up 2 (Week 24)
  The SF-36 is validated as a QoL measurement in the chronic pain population and is recommended by IMMPACT. Included here as an exploratory outcome with expected positive findings from pilot data collected by co-I Vasudev (unpublished) and other meditation interventions, which demonstrate moderate to large effect sizes. This measure is well-aligned to the intervention which is designed as a means of improving overall QoL more than as a disease treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Upshur, MD, Principal Investigator — Sinai Health System; Abhimanyu Sud, MD, Principal Investigator — Sinai Health System; Michelle Nelson, PhD, Principal Investigator — Sinai Health System
Locations (1):
- Bridgepoint Collaboratory, Sinai Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] MacCoon DG, Imel ZE, Rosenkranz MA, Sheftel JG, Weng HY, Sullivan JC, Bonus KA, Stoney CM, Salomons TV, Davidson RJ, Lutz A. The validation of an active control intervention for Mindfulness Based Stress Reduction (MBSR). Behav Res Ther. 2012 Jan;50(1):3-12. doi: 10.1016/j.brat.2011.10.011. Epub 2011 Nov 11. PMID 22137364
- [Background] MacCoon DG, MacLean KA, Davidson RJ, Saron CD, Lutz A. No sustained attention differences in a longitudinal randomized trial comparing mindfulness based stress reduction versus active control. PLoS One. 2014 Jun 23;9(6):e97551. doi: 10.1371/journal.pone.0097551. eCollection 2014. PMID 24955584
- [Background] Rayner L, Hotopf M, Petkova H, Matcham F, Simpson A, McCracken LM. Depression in patients with chronic pain attending a specialised pain treatment centre: prevalence and impact on health care costs. Pain. 2016 Jul;157(7):1472-9. doi: 10.1097/j.pain.0000000000000542. PMID 26963849
- [Background] McMillan D, Gilbody S, Richards D. Defining successful treatment outcome in depression using the PHQ-9: a comparison of methods. J Affect Disord. 2010 Dec;127(1-3):122-9. doi: 10.1016/j.jad.2010.04.030. Epub 2010 May 31. PMID 20569992
- [Background] Meader N, Mitchell AJ, Chew-Graham C, Goldberg D, Rizzo M, Bird V, Kessler D, Packham J, Haddad M, Pilling S. Case identification of depression in patients with chronic physical health problems: a diagnostic accuracy meta-analysis of 113 studies. Br J Gen Pract. 2011 Dec;61(593):e808-20. doi: 10.3399/bjgp11X613151. PMID 22137418
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Cunningham JL, Evans MM, King SM, Gehin JM, Loukianova LL. Opioid Tapering in Fibromyalgia Patients: Experience from an Interdisciplinary Pain Rehabilitation Program. Pain Med. 2016 Sep;17(9):1676-85. doi: 10.1093/pm/pnv079. Epub 2016 Jan 11. PMID 26755658
- [Background] Elliott TE, Renier CM, Palcher JA. Chronic pain, depression, and quality of life: correlations and predictive value of the SF-36. Pain Med. 2003 Dec;4(4):331-9. doi: 10.1111/j.1526-4637.2003.03040.x. PMID 14750909
- [Background] Hilton L, Hempel S, Ewing BA, Apaydin E, Xenakis L, Newberry S, Colaiaco B, Maher AR, Shanman RM, Sorbero ME, Maglione MA. Mindfulness Meditation for Chronic Pain: Systematic Review and Meta-analysis. Ann Behav Med. 2017 Apr;51(2):199-213. doi: 10.1007/s12160-016-9844-2. PMID 27658913
- [Derived] Cheng DK, Simpson R, Moineddin R, Katz J, Mulsant BH, Vasudev A, Greiver M, Hosseiny F, Inzitari M, Newman RI, Rivlin L, Foat KD, Furlan AD, Flannery JF, Telner D, Bosma R, Naimer M, Chung C, Pinto AD, Nelson MLA, Upshur R, Sud A. A Multi-Site, Randomized, Parallel-Group, Controlled Trial of Virtually-Delivered Sahaj Samadhi Meditation for the Management of Moderate Depressive Symptoms in Chronic Pain. J Pain Res. 2025 Jun 13;18:2925-2946. doi: 10.2147/JPR.S515229. eCollection 2025. PMID 40534615
- [Derived] Sud A, Nelson MLA, Cheng DK, Armas A, Foat K, Greiver M, Hosseiny F, Katz J, Moineddin R, Mulsant BH, Newman RI, Rivlin L, Vasudev A, Upshur R. Sahaj Samadhi Meditation versus a Health Enhancement Program for depression in chronic pain: protocol for a randomized controlled trial and implementation evaluation. Trials. 2020 Apr 7;21(1):319. doi: 10.1186/s13063-020-04243-z. PMID 32264945